CLINICAL TRIAL: NCT02900105
Title: Effect of Letrozole on Seminal Parameters in Men With Non Obstructive Azoospermia and Severe Oligozoospermia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Liu Shuling, Associate Consultant, KK Women's and Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014/123/D
Record Dates: First submitted 2016-08-30; First posted 2016-09-14 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Azoospermia, Nonobstructive; Oligozoospermia
MeSH Terms: conditions — Azoospermia, Nonobstructive; Oligospermia | interventions — Letrozole

ARMS (1):
- Letrozole (Experimental): Participants will be assigned to receive Letrozole 2.5 mg once a day for 4 months
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole — Letrozole 2.5mg (1 tablet) once a day for 4 months

SUMMARY:
The investigators hope to learn if Letrozole is effective and safe in improving severe male infertility by increasing testosterone, decreasing oestradiol and stimulating sperm production thereby improving sperm motility (movement) and concentration. The study is being conducted because Letrozole is not yet proven to be a standard treatment in subjects with absent or very low sperm counts. The investigators are hoping to determine whether Letrozole is equal or superior to no treatment.

DETAILED DESCRIPTION:
This is a pilot study with recruitment carried out in a single centre where participants will be assigned to receive Letrozole 2.5 mg once a day for 4 months. The following data will be collected: semen analyses, clinical history including smoking status, BMI, Y microdeletion, karyotype and FSH, LH, testosterone, E2, drug side effects and effects on libido. The following assessments will be performed before and 4 months after drug administration: sperm analyses, FSH, LH, E2 and testosterone measurements.

Prior to recruitment, the study participant would have undergone the routine investigations for evaluating azoospermia or severe oligozoospermia. These would include FSH, LH, testosterone, karyotyping, Y chromosome microdeletion genetic studies and at least 1 seminal analysis. Despite the availability of biochemical techniques to differentiate non-obstructive azoospermia (NOA) patients from obstructive azoospermia patients, fine needle aspiration (FNA) has been regarded as a highly informative and a minimally invasive method often routinely done in the investigation of azoospermia. All patients with NOA would have a FNA performed as part of their routine workup which would be done before recruitment and initiation of Letrozole. The safety of FNA use is also regarded as being supportive for the researchers against any possible patient lawsuits resulting from any impaired spermatogenesis induced by an off-label prescription. All oligozoospermic patients will be offered to have their sperm cryopreserved before drug administration. The investigations must have been performed within a 6 month time frame prior to recruitment.

There will be 3 clinic visits during the dosing period and 1 post dosing follow up visit. During the initial visit where recruitment into the study occurs, the participant will be prescribed the medication. One week later, a telephone interview will be conducted to review for side effects and arrange an early appointment at patient request. One month later, the participant will be reviewed in clinic and a side effect check list will be conducted. Telephone interviews will be conducted again at 2nd and 3rd month from administration of the drug. At 4th month from administration of the drug, the blood tests and semen analysis will be performed. It is likely that the participant will still be followed up for enrolment into IVF / ICSI programme should spontaneous pregnancy fail to occur. The window period for all clinic visits and telephone interviews is +/- 5 days.

ELIGIBILITY:
Inclusion Criteria

* Patients with non-obstructive azoospermia (absence of sperm in the pellets of two centrifuged semen samples collected 30-60 days apart)
* Patients with non-obstructive azoospermia who do not yield spermatozoa with fine needle aspiration (FNA)
* Patients with severe oligozoospermia (presence of sperm concentration less than 5 million per ml in both semen samples collected 30-60 days apart)
* Normal sperm appearance, consistency, liquefaction, volume and pH
* Patient must not possess any chromosomal aberrations

Exclusion Criteria

* Possible etiology of infertility present
* Seminal white blood cell concentration more than 10 million per ml
* Positive seminal culture analysis
* Positive urethral swab for chlamydia test
* Smoker
* Drug or alcohol abuse
* Ongoing medical treatment (gonadotropins, anabolic steroids, cancer chemotherapy, non-steroidal anti-inflammatory drugs, previous cancer radiotherapy or chemotherapy)
* Palpable varicocele
* X-ray exposure in the previous 8 months
* Y chromosome microdeletion
* Karyotype abnormalities (Klinefelter syndrome)

Ages: 21 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Sperm density | After 4 months dosage of Letrozole
Sperm motility | After 4 months dosage of Letrozole

SECONDARY OUTCOMES:
Total serum Testosterone level | After 4 months dosage of Letrozole
Total serum Estradiol level | After 4 months dosage of Letrozole
Total serum Follicle Stimulating Hormone level | After 4 months dosage of Letrozole
Total serum Luteinizing Hormone level | After 4 months dosage of Letrozole

CONTACTS AND LOCATIONS:
Overall Officials: Shuling Liu, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore